CLINICAL TRIAL: NCT05468905
Title: China Longitudinal Aging and Cognitive Impairment Study
Acronym: CLACIS
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Central Hospital of Lishui City (Other); Zhejiang Rehabilitation Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: wulab-CLACIS
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Aging; Mild Cognitive Impairment; Alzheimer Disease; Neurodegeneration
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum retention in -80℃ fridge for ApoE4 gene test etc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cognitive normal Aging (CN): Normal aging subjects with normal cognitive function
  Interventions: Other: None of intervention
- Subjective cognitive impairment (SCI): Self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event. Answering "yes" to both of the following questions: "Do you feel like your memory or thinking is becoming worse?" and "Does this concern you?"
  Interventions: Other: None of intervention
- Mild cognitive impairment (MCI): Mild cognitive impairment subjects with memory loss as predominant symptom
  Interventions: Other: None of intervention
- Alzheimer's disease (AD): Mild to moderate sporadic and familial Alzheimer disease subjects
  Interventions: Other: None of intervention
- Vascular cognitive impairment (VCI): Cognitive impairment subjects caused by cerebral vessel disease
  Interventions: Other: None of intervention

INTERVENTIONS:
Other: None of intervention — None of intervention

SUMMARY:
This is a multi-center longitudinal study that consists of five cohorts: cognitive normal aging (CN), Subjective cognitive impairment (SCI), mild cognitive impairment (MCI), Alzheimer's disease (AD) and vascular cognitive impairment (VCI). The goals of this study are as follow: 1.To establish longitudinal cohort study database containing comprehensive epidemiological data, neuropsychological test data, laboratory parameters, image data and biological samples. 2. To determine the risk factors of AD and other dementias. 3. To explore the conversion rates from CN to SCI, MCI or AD and the risk factors as well as biomarkers for the progression from CN to SCI, MCI or AD. 4. To explore and validate blood, CSF, urine, imaging and other biomarkers for the early detection and progression of AD.

DETAILED DESCRIPTION:
As the population ages in China, the number of patients with neurocognitive disorders such as Alzheimer's disease (AD) and vascular cognitive impairment (VCI) is steadily increasing. The burden of cognitive impairment in China has been an important public health problem. Cohort study on aging and cognitive impairment is urgent to better understand and address this issue. Early prevention, diagnosis and treatment are critical for reduction the burden of cognitive impairment. In this prospective study, subjects will be recruited into one of the five groups based on inclusion and exclusion criteria: 1) CN, 2) MCI 3) AD and 4) VCI. Each of the subjects will be followed up at designated time points up to 5 years. Epidemiological data, medical, imaging (MRI and PET scans), genetic information and various biological samples will be collected during the baseline and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Cognitive normal aging (CN) 1. 40 years and older , without cognitive impairment, MMSE≥22 2. Informed consent is signed by the participant
2. Subjective cognitive impairment (SCI) Participants aged 40 and older, with absence of dementia (by DSM IV and DSM V) criteria. Normal age-, sex-, and education-adjusted performance on standardized cognitive tests, which are used to classify mild cognitive impairment (MCI) or prodromal AD. Self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event. Answering "yes" to both of the following questions: "Do you feel like your memory or thinking is becoming worse?" and "Does this concern you?"
3. Mild cognitive impairment (MCI) 1. 40 years and older 2. Diagnosis according to 2004 Peterson's MCI criteria. 3. Clinical Dementia Rating (CDR) = 0.5. 4. Memory loss is prominent, and may also be with other cognitive domain impairment.

   5. Insidious onset, slow progress.
4. Alzheimer's disease (AD)

   1. 50 years and older
   2. Dementia is diagnosed according to the criteria described by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-R). The diagnosis of AD according to the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS- ADRDA) or National Institute on Aging and the Alzheimer's Assocation (NIA-AA) criteria.
   3. Subjects and their informed persons can complete relevant and follow-up examinations.
   4. Subjects or their authorized legal guardians sign the informed consent. Vascular cognitive impairment (VCI)

   1. 40 years and older 2. Diagnosis according to the criteria for small vessel VCI, with the following three core elements:

   1) Cognitive impairment: memory decline can be highlighted 2) Vascular factors 3) Causal relationship between cognitive impairment and vascular factors 3.Cognitive impairment lasts for 3 months or more, and the CDR global score ≥0.5 point.

   4. All patients need to meet the following MRI criteria:
   1. Multiple (≥3) small infarcts (3-20 mm in diameter) with or without any degree of white matter lesions (WML); or moderate to severe WML (Fazekas score ≥ 2) , with or without small infarction; or ≥ 1 small infarct in key parts of the cortex, such as: caudate nucleus, globus pallidus, thalamus et al.
   2. No WML caused by cortical infarction, watershed infarction, hemorrhage, hydrocephalus, or other causes (such as multiple sclerosis).
   3. No hippocampus or entorhinal cortex atrophy, Medial Temporal Lobe Atrophy (MTA)≤ 1 point.

   5. Subjects and their informed persons can complete relevant and follow-up examinations.

   6. Subjects or their authorized legal guardians sign the informed consent.

   Exclusion Criteria:

   Cognitive normal aging (CN)
   1. any disease that can cause cognitive impairment (such as Alzheimer's disease, dementia with Lewy bodies (DLB), frontotemporal dementia (FTLD), Parkinson's disease dementia (PDD), intracranial masses that impair cognition, history of severe brain trauma, normal pressure hydrocephalus, cerebrovascular disease with obvious clinical symptoms, etc.
   2. sequelae after previous history of severe central nervous system infection, multiple sclerosis, autoimmune encephalitis, Hashimoto's encephalopathy, etc.
   3. previous history of instable epilepsy
   4. systemic diseases affect the central nervous system, for abnormal liver and kidney functions (abdominal dialysis, hemodialysis, AST≥3× upper limit of normal value (ULN), ALT≥3× upper limit of normal value (ULN) or total bilirubin ≥2×ULN
   5. history of hereditary diseases that affect cognitive function (such as Huntington's disease, down syndrome, CADASIL, adrenal leukodystrophy, mitochondrial encephalopathy, etc.)
   6. long-term heavy drinking history (alcohol content more than 42 degree liquor, more than 150g/day, alcohol consumption more than 12 months)
   7. history of severe pulmonary diseases (COPD, pulmonary encephalopathy)
   8. history of serious cardiovascular disease (heart failure, severe hypertension)
   9. infection and immune-related diseases affecting the central nervous system (systemic lupus erythematosus, undertreated HIV infection or a history of CNS syphilis infection, etc.)
   10. metabolic and endocrine disorders (requiring new treatment or adjustment of current treatment for thyroid dysfunction, folate or vitamin B12 deficiency)
   11. unstable psychosis or long-term use of antipsychotic drugs (more than 6 months)
   12. history of malignant tumors (tumors of nervous system and other sites) active for nearly 1 year
   13. contraindications for MRI (e.g. pacemakers, stents, claustrophobia, etc.) or do not cooperate or cannot carry out PET examination
   14. uneducated illiterates
   15. hearing impairment, visual impairment and poor coordination
   16. withdraw or reject the study Subjective cognitive impairment (SCI) and Mild cognitive impairment (MCI)

   <!-- -->

   1. With history of stroke and a neurological focal sign, the imaging findings are consistent with cerebral vascular disease (Fazekas score ≥ 2 points).
   2. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
   3. Other systemic diseases that can cause cognitive impairment（such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.）.
   4. Mental and neurodevelopmental retardation.
   5. Other diseases known to cause cognitive impairment.
   6. Contraindications to nuclear magnetics.
   7. Suffering from a disease that cannot be combined with cognitive examination.
   8. Refuse to draw blood.
   9. Refuse to sign the informed consent at baseline Alzheimer's disease (AD)

   <!-- -->

   1. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
   2. Other systemic diseases that can cause cognitive impairment（such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.）.
   3. Mental and neurodevelopmental retardation.
   4. Other diseases known to cause cognitive impairment.
   5. Contraindications to nuclear magnetics.
   6. Suffering from a disease that cannot be combined with cognitive examination.
   7. Refuse to draw blood.
   8. Refuse to sign the informed consent at baseline Vascular cognitive impairment (VCI)

   <!-- -->

   1. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.).
   2. Other systemic diseases that can cause cognitive impairment（such as liver, renal, and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.）.
   3. Other diseases known to cause cognitive impairment.
   4. Hereditary or inflammatory small vessel disease, such as cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL).
   5. Contraindications to nuclear magnetics.
   6. Refuse to draw blood.
   7. Refuse to sign the informed consent at baseline

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female participants ages 40 to 99 years
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence, incidence of cognitive impairment caused by neurological disease such as AD, VCI and other types of dementia | 5 years
  All of the participants will be evaluated by cognitive assessment scale annually.
The conversion rate of normal aging to SCI, MCI and AD | 5 years
  All of the participants will be evaluated by cognitive assessment scale annually.
The fluid biomarkers for normal aging, SCI, MCI and AD diagnosis | 5 years
  Cerebrospinal fluid, plasma, saliva and urine biomarkers included Aβ42, Aβ40, phosphated tau and total tau, and other novel biomarkers.
The imaging biomarkers for normal aging, MCI and AD diagnosis | 5 years
  Imaging biomarkers included cerebral atrophy, amyloid and tau deposition of whole brain or hippocampus, glucose metabolism and other novel biomarkers.
Gut microbiota | 5 years
  Fecal microbiome will be analyzed by 16S rRNA gene sequencing and metagenome sequencing.
Gait | 5 years
  Gait characteristics such as stride-to-stride variability of stride time, and gait speed were evaluated by 3D gait detection.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ying Wu, M.D&Ph.D, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (2):
- China (2):
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Lishui central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No